CLINICAL TRIAL: NCT01283399
Title: A Non-interventional Multicenter Study of MabThera® (Rituximab) in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: An Observational Study of Rituximab in Combination With Methotrexate in Participants With Active Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25270
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rituximab + Methotrexate: All participants with active refractory RA who were eligible to receive treatment with methotrexate and rituximab in the Investigators' opinion as per the routine clinical practice following inadequate response to a single cycle of anti-TNF therapy.

SUMMARY:
This observational study will assess the efficacy and safety of combination of rituximab (MabThera) and methotrexate in participants with active refractory rheumatoid arthritis (RA) who have failed to respond to a single course of anti-tumor necrosis factor (TNF) therapy in routine clinical practice. Data will be collected from participants for 12 months after the first dose of rituximab or a minimum of 6 months following a rituximab re-treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis
* Inadequate response to a single TNF inhibitor
* Participants receiving rituximab therapy in accordance with the prescribing information
* Signed data release form within 6 weeks (42 days) of initiating rituximab therapy
* Women of childbearing potential must use effective form of contraception

Exclusion Criteria:

* Contra-indication to receive rituximab according to the local labelling
* Previous treatment with rituximab
* Treatment with any investigational drug within 30 days prior to enrolment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants with active refractory RA who were eligible to receive treatment with methotrexate and rituximab in the Investigators' opinion as per the routine clinical practice following inadequate response to a single cycle of anti-TNF therapy.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score Based on 28-joints Count (DAS28) | Up to 5 years

SECONDARY OUTCOMES:
Reasons for Re-treatment With Rituximab Within 6 Months of the First Treatment | Up to 5 years
Disease Activity Score Based on 28-joints Count (DAS28) 6 Months After the Re-treatment With Rituximab | 6 Months After the Re-treatment With Rituximab (up to 5 years)
Demographics of Participants Eligible to Receive Rituximab | Baseline
Number of Participants With Adverse Events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Lebanon (3):
  - Beirut
  - Byblos
  - Tripoli